CLINICAL TRIAL: NCT02854436
Title: A Phase 2 Efficacy and Safety Study of Niraparib in Men With Metastatic Castration-Resistant Prostate Cancer and DNA-Repair Anomalies
Brief Title: An Efficacy and Safety Study of Niraparib in Men With Metastatic Castration-Resistant Prostate Cancer and DNA-Repair Anomalies
Acronym: Galahad
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108208; 64091742PCR2001 (Other: Janssen Research & Development, LLC); 2016-002057-38 (EudraCT Number)
Record Dates: First submitted 2016-08-01; First posted 2016-08-03 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate cancer; CRPC; Metastatic castrate-resistant prostate cancer; Prostate neoplasm; Galahad; Niraparib; DNA anomalies; DNA defect; PARP inhibitor; PARPi
MeSH Terms: conditions — Prostatic Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Niraparib (Experimental): Participants will receive 300 milligram (mg) niraparib (3 capsules*100 mg) orally once daily.
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Participants will receive 300 mg niraparib (3 capsules*100 mg) orally once daily.
  Other Names: JNJ-64091742

SUMMARY:
The purpose of this study is to assess the efficacy, safety, and pharmacokinetics of niraparib in men with metastatic castration-resistant prostate cancer (mCRPC) and deoxyribonucleic acid (DNA) repair anomalies.

DETAILED DESCRIPTION:
This is a multicenter and open-label (participants and researchers are aware of the treatment that participants are receiving) study that consists of 4 phases: a Prescreening Phase for biomarker evaluation only, a Screening Phase, a Treatment Phase (Cycle 1 Day 1 and will continue until the study drug is discontinued), a Follow-up Phase (every 3 months after end of treatment visit), and a Long-term Extension Phase (until participants no longer derive benefit from treatment or until further notification on different means of study treatment). Participants will be monitored for safety during the study period, and up to 30 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer (mixed histology is acceptable, with the exception of the small cell pure phenotype, which is excluded)
* Received a taxane-based chemotherapy for the treatment of metastatic prostate cancer with evidence of disease progression on or after treatment, or discontinued from a taxane-based chemotherapy due to an adverse event
* Received a second-generation or later androgen receptor (AR)-targeted therapy (for example, abiraterone acetate plus prednisone, enzalutamide, apalutamide) for the treatment of metastatic prostate cancer with evidence of disease progression or non-metastatic castration-resistant prostate cancer with evidence of subsequent metastasis
* Biomarker-positive by at least one of the following criteria: (a) Biallelic deoxyribonucleic acid (DNA)-repair anomaly based on a sponsor validated blood or tissue assay; (b) Germline pathogenic Breast Cancer gene (BRCA) 1 or BRCA2 by any test (somatic local results must be confirmed as positive by the sponsor-validated assay before dosing)
* Progression of metastatic prostate cancer in the setting of castrate levels of testosterone or history of bilateral orchiectomy at study entry

Exclusion Criteria:

* Prior treatment with a poly (adenosine diphosphate [ADP] ribose) polymerase (PARP) inhibitor
* Prior platinum-based chemotherapy for the treatment of prostate cancer
* Known history or current diagnosis of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)
* Symptomatic or impending cord compression
* Symptomatic brain metastases

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2016-08-31 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2023-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (110):
- United States (23):
  - Tucson, Arizona
  - Los Angeles, California
  - Riverside, California
  - Sacramento, California
  - Aurora, Colorado
  - Denver, Colorado
  - Evanston, Illinois
  - Danville, Kentucky
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Omaha, Nebraska
  - New York, New York
  - Durham, North Carolina
  - Lancaster, Pennsylvania
  - Philadelphia, Pennsylvania
  - Myrtle Beach, South Carolina
  - Houston, Texas
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Seattle, Washington
  - Madison, Wisconsin
- Australia (10):
  - Camperdown
  - Darlinghurst
  - East Albury
  - Kurralta Park
  - Macquarie University
  - Melbourne
  - Murdoch
  - Port Macquarie
  - Randwick
  - Wahroonga
- Belgium (11):
  - Aalst
  - Brussels
  - Charleroi
  - Ghent
  - Haine-Saint-Paul
  - Hasselt
  - Kortrijk
  - Liège
  - Namur
  - Ottignies
  - Wilrijk
- Brazil (10):
  - Barretos
  - Belo Horizonte
  - Curitiba
  - Fortaleza
  - Ijuí
  - Itajaí
  - Joinville
  - Natal
  - Salvador
  - São Paulo
- Canada (5):
  - Vancouver, British Columbia
  - Oshawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- Denmark (4):
  - Aarhus N
  - Copenhagen N
  - Herlev
  - Odense C
- France (9):
  - Avignon
  - Besançon
  - Caen
  - Lyon
  - Nice
  - Paris
  - Reims
  - Strasbourg
  - Villejuif
- Israel (5):
  - Beersheba
  - Haifa
  - Kfar Saba
  - Ramat Gan
  - Zrifin
- Netherlands (5):
  - Alkmaar
  - Amsterdam
  - Groningen
  - Maastricht
  - Rotterdam
- Russia (3):
  - Moscow
  - Omsk
  - Tomsk
- Seoul, South Korea
- Spain (9):
  - Barcelona
  - Córdoba
  - Madrid
  - Málaga
  - Pozuelo de Alarcón
  - Santander
  - Santiago de Compostela
  - Seville
  - Valencia
- Sweden (4):
  - Gothenburg
  - Lund
  - Stockholm
  - Umeå
- Taiwan (5):
  - Kaohsiung City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan
- United Kingdom (6):
  - Blackburn
  - Bristol
  - Cardiff
  - Exeter
  - London
  - Preston

REFERENCES:
- [Derived] Smith MR, Sandhu S, George DJ, Chi KN, Saad F, Thiery-Vuillemin A, Stahl O, Olmos D, Danila DC, Gafanov R, Castro E, Moon H, Joshua AM, Mason GE, Espina BM, Liu Y, Lopez-Gitlitz A, Francis P, Bevans KB, Fizazi K. Health-related quality of life in GALAHAD: A multicenter, open-label, phase 2 study of niraparib for patients with metastatic castration-resistant prostate cancer and DNA-repair gene defects. J Manag Care Spec Pharm. 2023 Jul;29(7):758-768. doi: 10.18553/jmcp.2023.29.7.758. PMID 37404070
- [Derived] Smith MR, Scher HI, Sandhu S, Efstathiou E, Lara PN Jr, Yu EY, George DJ, Chi KN, Saad F, Stahl O, Olmos D, Danila DC, Mason GE, Espina BM, Zhao X, Urtishak KA, Francis P, Lopez-Gitlitz A, Fizazi K; GALAHAD investigators. Niraparib in patients with metastatic castration-resistant prostate cancer and DNA repair gene defects (GALAHAD): a multicentre, open-label, phase 2 trial. Lancet Oncol. 2022 Mar;23(3):362-373. doi: 10.1016/S1470-2045(21)00757-9. Epub 2022 Feb 4. PMID 35131040

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For long-term extension (LTE) phase, as pre planned in the protocol no efficacy analysis was performed. Due to change in the conduct of the study, no adverse events data were collected and thus no adverse event data were reported for the LTE phase.
Groups:
- Niraparib: Male Subjects who were over the age of 18 years with metastatic castration-resistant prostate cancer (based (mCRPC) and deoxyribonucleic acid (DNA) repair anomalies and who had received prior taxane-based chemotherapy milligrams chemotherapy and androgen receptor (AR)-targeted therapy received once daily oral dose of 300 milligrams (or(mg) niraparib capsules starting Day 1 until disease progression, unacceptable toxicity, death, or termination subjects termination of the study by the sponsor (up to 52 months). After completion of treatment phase, subjects were offered entry into the long-term extension (LTE) phase (which was planned as per protocol amendment 8, dated 17-Jul-2020) with a separate informed consent and to continue treatment per the investigator's discretion until no benefits from treatment or Sponsor's decision.
Period: Overall Study
Arm/Group | Niraparib
Started | 289
Intent to Treat Participants (Breast Cancer Gene [BRCA] and Non-BRCA Participants) | 223 (There were 142 BRCA participants and 81 non-BRCA participants.)
Completed | 0
Not Completed | 289
Not completed — Adverse Event | 1
Not completed — Death | 208
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 24
Not completed — Other | 45
Not completed — Physician Decision | 6

BASELINE CHARACTERISTICS:
Arm/Group | Niraparib
Number analyzed (Participants) | 289
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 289
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 16
  Black or African American | 9
  Native Hawaiian or Other Pacific Islander | 0
  White | 205
  More than one race | 3
  Unknown or Not Reported | 51
  Other | 5
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRALIA | 31
  BELGIUM | 18
  BRAZIL | 12
  CANADA | 21
  DENMARK | 1
  FRANCE | 48
  ISRAEL | 6
  NETHERLANDS | 6
  RUSSIAN FEDERATION | 7
  SOUTH KOREA | 5
  SPAIN | 39
  SWEDEN | 24
  TAIWAN | 9
  UNITED KINGDOM | 17
  UNITED STATES | 45

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) for Participants With Measurable Metastatic Castration-resistant Prostate Cancer (mCRPC) and Breast Cancer Gene (BRCA) Mutation
Description: ORR defined as percentage of participants with BRCA DNA-repair anomalies and measurable disease whose best response is either complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) and with no evidence of bone progression per Prostate Cancer Working Group 3 (PCWG3) criteria.
Time Frame: Up to 52 months
Population: Measurable intent to treat (ITT) population also referred to as efficacy analysis set included all participants who received at least 1 dose of study drug and have BRCA (biallelic or germline DNA-repair anomalies) and measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Niraparib
Number analyzed (Participants) | 76
percentage of participants | 34.2 [23.7 to 46.0]

2. Secondary Outcome: Objective Response Rate for Participants With Measurable Metastatic Castration-resistant Prostate Cancer (mCRPC) and Non-Breast Cancer Gene (BRCA) Mutation
Description: ORR defined as percentage of participants with BRCA deoxyribonucleic acid (DNA)-repair anomalies and measurable disease whose best response is either CR or PR per RECIST 1.1 and with no evidence of bone progression per PCWG3 criteria.
Time Frame: Up to 52 months
Population: Measurable ITT analysis set included all participants who received at least 1 dose of study drug and have non-BRCA (biallelic DNA-repair anomaly) and measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Niraparib
Number analyzed (Participants) | 47
percentage of participants | 10.6 [3.5 to 23.1]

3. Secondary Outcome: Circulating Tumor Cells (CTC) Response Rate
Description: CTC response rate was defined as the percentage of participants with CTC equals to (=) 0 per 7.5 milliliter (mL) blood at 8 weeks post-baseline in participants with baseline CTC greater than (>) 0.
Time Frame: At 8 weeks post-baseline
Population: ITT analysis set included all participants who received at least 1 dose of study drug. Here 'N' (number of participants analysed) specifies the participants with baseline CTC (per 7.5 mL blood) > 0. Here, 'n' (number analyzed) specifies the number of participants evaluated for specific categories.
Measure: Number; unit: percentage of participants
Arm/Group | Niraparib
Number analyzed (Participants) | 202
percentage of participants
  BRCA: number analyzed (Participants) | 131
  BRCA | 23.7
  Non-BRCA: number analyzed (Participants) | 71
  Non-BRCA | 8.5

4. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from enrollment to death from any cause.
Time Frame: Up to 52 months
Population: ITT analysis set included participants who had received at least 1 dose of study drug. Here, 'n' (number analyzed) specifies the number of participants evaluated for specific categories.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib
Number analyzed (Participants) | 223
months
  BRCA: number analyzed (Participants) | 142
  BRCA | 13.01 [11.04 to 14.29]
  Non-BRCA: number analyzed (Participants) | 81
  Non-BRCA | 9.63 [8.05 to 13.44]

5. Secondary Outcome: Radiographic Progression-Free Survival (rPFS)
Description: rPFS was defined as time from enrollment to radiographic progression or death from any cause, whichever occurred first. Radiographic progression was evaluated per RECIST 1.1 criteria for soft tissue disease and per PCWG3 criteria for bone disease.
Time Frame: Up to 52 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib
Number analyzed (Participants) | 223
months
  BRCA: number analyzed (Participants) | 142
  BRCA | 8.08 [5.55 to 8.38]
  Non-BRCA: number analyzed (Participants) | 81
  Non-BRCA | 3.71 [1.97 to 5.49]

6. Secondary Outcome: Time to Radiographic Progression
Description: Time to radiographic progression is defined as time from enrollment to radiographic progression or death due to disease progression, whichever occurs first. Disease progression is defined as at least a 20 percent (%) increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: Up to 52 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib
Number analyzed (Participants) | 223
months
  BRCA: number analyzed (Participants) | 142
  BRCA | 8.08 [5.75 to 8.97]
  Non-BRCA: number analyzed (Participants) | 81
  Non-BRCA | 3.78 [2.00 to 5.55]

7. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Progression
Description: Time to PSA progression was defined as time from enrollment to the first date of documented PSA progression based on PCWG3 criteria. A participant was considered to have a PSA progression if the PSA level had a 25 percent (%) or greater increase from nadir and an absolute increase of 2 nanograms per milliliter (ng/mL) or more, which is confirmed by a second value obtained in 3 or more weeks.
Time Frame: Up to 52 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib
Number analyzed (Participants) | 223
months
  BRCA: number analyzed (Participants) | 142
  BRCA | 5.13 [4.60 to 5.59]
  Non-BRCA: number analyzed (Participants) | 81
  Non-BRCA | 3.65 [2.83 to 3.71]

8. Secondary Outcome: Time to Symptomatic Skeletal Event (SSE)
Description: Time to SSE was defined as the time from enrollment to first occurrence of one of the following symptomatic skeletal events: tumor-related spinal cord compression, radiation to bone to relieve skeletal symptoms, surgery to bone or need for tumor-related orthopedic surgical intervention, symptomatic or pathologic fracture.
Time Frame: Up to 52 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib
Number analyzed (Participants) | 223
months
  BRCA: number analyzed (Participants) | 142
  BRCA | 13.80 [10.41 to NA] — Here, 'NA' indicates that upper limit of confidence interval was not estimable due to less number of events.
  Non-BRCA: number analyzed (Participants) | 81
  Non-BRCA | 10.35 [8.18 to NA] — Here, 'NA' indicates that upper limit of confidence interval was not estimable due to less number of events.

9. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response is defined as time from CR or PR to radiographic progression of disease, unequivocal clinical progression or death, whichever occurs first. Unequivocal clinical progression defined as one or more of following: 1) deterioration in Eastern Cooperative Oncology Group Performance Status (ECOG PS) to Grade 3 or higher; 2) need to initiate any of following because of tumor progression (even in absence of radiographic evidence of disease): alternative anticancer therapy for prostate cancer, radiation therapy, surgical interventions for complications due to tumor progression.
Time Frame: Up to 52 months
Population: Measurable ITT responder analysis set included all participants who received at least 1 dose of study drug, responded to it and have BRCA or non-BRCA and measurable disease at baseline. Here, 'n' (number analyzed) specifies the number of participants evaluated for specific categories.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Niraparib
Number analyzed (Participants) | 31
months
  BRCA: number analyzed (Participants) | 26
  BRCA | 5.55 [3.91 to 7.20]
  non-BRCA: number analyzed (Participants) | 5
  non-BRCA | 5.16 [2.14 to NA] — Here, 'NA' indicates that upper limit of confidence interval was not estimable due to less number of events.

10. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Time Frame: Up to 52 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib
Number analyzed (Participants) | 289
Participants | 288

11. Secondary Outcome: Number of Participants With Worst Toxicity Grades for Clinical Laboratory Tests Based on National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Description: Number of participants with worst toxicity grades for clinical laboratory tests (chemistry and hematology) based on NCI-CTCAE were reported. The chemistry laboratory parameters were: alanine aminotransferase (ALT) increased, alkaline phosphatase increased, aspartate aminotransferase (AST) increased, blood bilirubin increased, creatinine increased, gamma glutamyl transferase (GGT) increased and the hematology parameters were: hemoglobin increased, lymphocyte count increased. Grading was done as: Grade 1 (=mild), Grade 2 (=moderate), Grade 3 (=severe) and Grade 4 (=potentially life-threatening).
Time Frame: Up to 52 months
Population: Safety analysis set included all participants who received at least 1 dose of study drug and with at least one postbaseline assessment for the specific lab test within the time period. Here, 'n' (number analyzed) specifies the number of participants evaluated for specific categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Niraparib
Number analyzed (Participants) | 283
Participants
  ALT increased (Grade 1 or 2) | 67
  ALT increased (Grade 3 or 4) | 4
  Alkaline phosphatase increased (Grade 1 or 2) | 102
  Alkaline phosphatase increased (Grade 3 or 4) | 7
  AST increased (Grade 1 or 2) | 70
  AST increased (Grade 3 or 4) | 4
  Blood bilirubin increased (Grade 1 or 2) | 9
  Blood bilirubin increased (Grade 3 or 4) | 2
  Creatinine increased (Grade 1 or 2) | 45
  Creatinine increased (Grade 3 or 4) | 2
  GGT increased (Grade 1 or 2): number analyzed (Participants) | 282
  GGT increased (Grade 1 or 2) | 105
  GGT increased (Grade 3 or 4): number analyzed (Participants) | 282
  GGT increased (Grade 3 or 4) | 14
  Hemoglobin increased (Grade 1 or 2) | 0
  Hemoglobin increased (Grade 3 or 4) | 0
  Lymphocyte count increased (Grade 1 or 2) | 6
  Lymphocyte count increased (Grade 3 or 4) | 0

ADVERSE EVENTS:
Time Frame: Up to 52 months
Description: Safety analysis set included all participants who received at least 1 dose of study drug. Due to change in the conduct of the study, no adverse events data were collected and thus no adverse event data were reported for the LTE phase.
Arm/Group | Niraparib
All-Cause Mortality (participants affected / at risk) | 208/289
Serious Adverse Events (participants affected / at risk) | 134/289
Other Adverse Events (participants affected / at risk) | 280/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib (N=289)
Anaemia (Blood and lymphatic system disorders) | 13
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 17
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 4
Acute Abdomen (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Inflammatory Bowel Disease (Gastrointestinal disorders) | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 5
Rectal Haemorrhage (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Volvulus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 4
Facial Pain (General disorders) | 1
Fatigue (General disorders) | 4
General Physical Health Deterioration (General disorders) | 8
Non-Cardiac Chest Pain (General disorders) | 1
Pain (General disorders) | 2
Performance Status Decreased (General disorders) | 1
Pyrexia (General disorders) | 4
Systemic Inflammatory Response Syndrome (General disorders) | 1
Abdominal Infection (Infections and infestations) | 1
Abscess Jaw (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Escherichia Urinary Tract Infection (Infections and infestations) | 2
Herpes Zoster (Infections and infestations) | 1
Infected Lymphocele (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Malaria (Infections and infestations) | 1
Neutropenic Sepsis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 2
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pneumonia Haemophilus (Infections and infestations) | 1
Pyelonephritis Acute (Infections and infestations) | 2
Sepsis (Infections and infestations) | 5
Septic Shock (Infections and infestations) | 2
Skin Infection (Infections and infestations) | 1
Spinal Cord Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 3
Urosepsis (Infections and infestations) | 2
Cystitis Radiation (Injury, poisoning and procedural complications) | 1
Extradural Haematoma (Injury, poisoning and procedural complications) | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Hip Fracture (Injury, poisoning and procedural complications) | 2
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Blood Calcium Increased (Investigations) | 1
Blood Creatinine Increased (Investigations) | 1
Electrocardiogram QT Prolonged (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 7
Bone Pain (Musculoskeletal and connective tissue disorders) | 3
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastrointestinal Stromal Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered State of Consciousness (Nervous system disorders) | 1
Cauda Equina Syndrome (Nervous system disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Headache (Nervous system disorders) | 6
Ischaemic Stroke (Nervous system disorders) | 2
Monoparesis (Nervous system disorders) | 1
Nerve Compression (Nervous system disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Paraparesis (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Spinal Cord Compression (Nervous system disorders) | 6
Syncope (Nervous system disorders) | 2
Transient Ischaemic Attack (Nervous system disorders) | 1
Confusional State (Psychiatric disorders) | 2
Acute Kidney Injury (Renal and urinary disorders) | 2
Haematuria (Renal and urinary disorders) | 6
Renal Impairment (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 2
Prostatitis (Reproductive system and breast disorders) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Lung Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 1
Embolism (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Phlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Niraparib (N=289)
Anaemia (Blood and lymphatic system disorders) | 154
Leukopenia (Blood and lymphatic system disorders) | 27
Lymphopenia (Blood and lymphatic system disorders) | 24
Neutropenia (Blood and lymphatic system disorders) | 54
Thrombocytopenia (Blood and lymphatic system disorders) | 94
Abdominal Pain (Gastrointestinal disorders) | 23
Constipation (Gastrointestinal disorders) | 98
Diarrhoea (Gastrointestinal disorders) | 48
Dry Mouth (Gastrointestinal disorders) | 20
Dyspepsia (Gastrointestinal disorders) | 21
Nausea (Gastrointestinal disorders) | 167
Stomatitis (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 109
Asthenia (General disorders) | 45
Fatigue (General disorders) | 105
Oedema Peripheral (General disorders) | 41
Pyrexia (General disorders) | 17
Alanine Aminotransferase Increased (Investigations) | 17
Aspartate Aminotransferase Increased (Investigations) | 20
Blood Alkaline Phosphatase Increased (Investigations) | 26
Electrocardiogram QT Prolonged (Investigations) | 17
Gamma-Glutamyltransferase Increased (Investigations) | 25
Weight Decreased (Investigations) | 50
Decreased Appetite (Metabolism and nutrition disorders) | 93
Arthralgia (Musculoskeletal and connective tissue disorders) | 43
Back Pain (Musculoskeletal and connective tissue disorders) | 59
Bone Pain (Musculoskeletal and connective tissue disorders) | 30
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 29
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 30
Dizziness (Nervous system disorders) | 19
Dysgeusia (Nervous system disorders) | 17
Headache (Nervous system disorders) | 30
Insomnia (Psychiatric disorders) | 24
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39
Hot Flush (Vascular disorders) | 17
Hypertension (Vascular disorders) | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT02854436/Prot_002.pdf
  • Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT02854436/SAP_003.pdf